CLINICAL TRIAL: NCT05116410
Title: A Single- and Multiple-Ascending Dose Study in Healthy Subjects to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HS-20094
Brief Title: A Study of HS-20094 in Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HS-20094-101
Record Dates: First submitted 2021-10-29; First posted 2021-11-11 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2021-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HS-20094 (Single dose) (Experimental): Escalating doses of HS-20094 administered subcutaneously (SC) once in healthy participants.
  Interventions: Drug: HS-20094
- HS-20094 (Multiple doses) (Experimental): Escalating doses of HS-20094 administered SC once weekly for four weeks in healthy participants.
  Interventions: Drug: HS-20094
- Placebo (Single dose) (Placebo Comparator): Placebo administered SC once in healthy participants.
  Interventions: Drug: Placebo
- Placebo (Multiple doses) (Placebo Comparator): Placebo administered SC once weekly for four weeks in healthy participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HS-20094 — Administrated SC
  Other Names: HS-20094 injection
  Arms: HS-20094 (Multiple doses); HS-20094 (Single dose)
Drug: Placebo — Administrated SC
  Other Names: Placebo injection
  Arms: Placebo (Multiple doses); Placebo (Single dose)

SUMMARY:
This study includes two parts (Single Ascending Dose, SAD; Multiple-Ascending Dose, MAD) and enrolls healthy participants. Participants in SAD accept single subcutaneous (SC) injection of HS-20094 and participants in MAD accept SC injection of HS-20094 once weekly for 4 weeks. The main purpose of this study is to determine 1) The safety of HS-20094; 2) How much HS-20094 gets into the bloodstream and how long it takes the body to get rid of it.3) How HS-20094 affects the levels of blood sugar, insulin and weight.

ELIGIBILITY:
Inclusion Criteria:

1. Screening weight of male ≥50 kg, female≥45 kg and 19≤BMI≤28
2. Subjects agree to use an effective method of contraception and avoid sperm or egg donation for the duration of the study and for 6 months following the last dose of investigational product
3. Agree to avoid alcohol, foods and beverages containing xanthine or caffeine (including chocolate, tea, coffee, cola, etc.) from 48 hours prior to administration to last visit, and to avoid strenuous exercise

Exclusion Criteria:

1. Pregnant or lactating women
2. Subjects have a medical history of cardiovascular, respiratory, liver, kidney, digestive tract, mental, neurological, hematology or metabolic abnormalities (e.g., repeated hypoglycemia for unknown reasons) and are judged not suitable for this study by the investigator.
3. Subjects with abnormal screening vital signs, physical examination, laboratory examination or 12 lead electrocardiogram results with clinical significance
4. Have a history of drug allergy, or known allergies to HS-20094, glucagon-like peptide (GLP)-1 analogs, or glucose-dependent insulinotropic polypeptide (GIP) receptor agonism
5. Received systemic steroid therapy, immunomodulator therapy or chemotherapy in the 3 months prior to screening, or are likely to receive these treatments during the study period
6. Have a history of digestive disease (e.g., gastroesophageal reflux disease, gallbladder disease, or chronic enteritis) that may affect gastrointestinal adverse events assessment or any other gastrointestinal disease (e.g., gastric bypass surgery, pyloric stenosis, etc.) that may affect gastric emptying
7. Have a diet, weight loss treatment or significant lifestyle changes prior to 30 days of administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse event (AE), serious adverse event (SAE), AE leading to study discontinuation, AE severity and relation with study drug | Time of Inform Consent Form to Day 29 (SAD) or Day 50 (MAD)
  A summary of AEs and SAEs, AE leading to study discontinuation, AE severity and relation with study drug will be reported in the reported adverse events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Cmax of HS-20094 | Baseline to Day 22 (SAD) or Day 43 (MAD)
  PK: Cmax of HS-20094
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of HS-20094 | Baseline to Day 22 (SAD) or Day 43 (MAD)
  PK: AUC of HS-20094
Pharmacokinetics (PK): Tmax of HS-20094 | Baseline to Day 22 (SAD) or Day 43 (MAD)
  PK: Tmax of HS-20094
Pharmacodynamics (PD): AUC of glucose | Day 22 (MAD)
  PD: AUC of glucose
Pharmacodynamics (PD): AUC of insulin | Day 22 (MAD)
  PD: AUC of insulin
Weight change | baseline to Day 29 (SAD) or Day 50 (MAD)

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Cui, Principal Investigator — Beijing University First Hospital
Locations (1):
- Beijing University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No